CLINICAL TRIAL: NCT02963298
Title: Pilot Trial Concerning Glutamate Elimination With CRRT for Neurological Outcome After Cardiac Arrest
Brief Title: CRRT for Glutamate Elimination After Cardiac Arrest
Acronym: GCRRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. Storm (Other)
Responsible Party: Sponsor-Investigator, C. Storm, PD Dr. med., Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Glu2016
Record Dates: First submitted 2016-10-11; First posted 2016-11-15 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Reperfusion Syndrome
MeSH Terms: interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CRRT after cardiac arrest (Active Comparator): Continuous renal replacement therapy (CRRT) after cardiac arrest for 72 hours for elimination of Glutamate. Repetitive testing of blood Glutamate levels.
  Interventions: Procedure: Continuous renal replacement therapy
- control (No Intervention): Repetitive testing of blood Glutamate levels without CRRT

INTERVENTIONS:
Procedure: Continuous renal replacement therapy
  Arms: CRRT after cardiac arrest

SUMMARY:
Glutamate is known to be a mediator for apoptosis after brain hypoxia e.g. due to cardiac arrest. This pilot trial evaluates the possibility of elimination of Glutamate by CRRT after cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* post cardiac arrest

Exclusion Criteria:

* hemodynamic instable
* in-hospital cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Glutamate blood concentration in intervention arm over the time | 72 hours
  Reduction of blood Glutamate concentration by renal replacement therapy

SECONDARY OUTCOMES:
number of participants with abnormal outcome parameters | up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Christian Storm, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Derived] Nee J, Jorres A, Krannich A, Leithner C, Schroeder T, Munk AL, Enghard P, Moore C, Steppan S, Storm C. Elimination of glutamate using CRRT for 72 h in patients with post-cardiac arrest syndrome: A randomized clinical pilot trial. Resuscitation. 2019 Nov;144:54-59. doi: 10.1016/j.resuscitation.2019.09.020. Epub 2019 Sep 23. PMID 31557520